CLINICAL TRIAL: NCT01235169
Title: Evaluation of the Proximal Femoral Nail Antirotation With Cement Augmentation in Osteoporotic Femoral Neck Fractures
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: WEIL02-HMO-CTIL
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Proximal Femur Fracture
MeSH Terms: conditions — Proximal Femoral Fractures

ARMS (1):
- Proximal Femoral Nail Antirotation (Experimental): Proximal Femoral Nail Antirotation(PFNA) with cement augmentation
  Interventions: Device: Proximal Femoral Nail Antirotation(PFNA) with cement augmentation

INTERVENTIONS:
Device: Proximal Femoral Nail Antirotation(PFNA) with cement augmentation

SUMMARY:
This is an open multicenter study, evaluating a new operative technique in femur neck fractures. The treatment consist of augmentated nails in cases of subtrochanteric or inter fracture due to osteoporosis.There two routine surgical techniques in femoral neck fractures:

1. Insertion an intramedullary nail (without augmentation) to the bone.
2. insertion a nail and metal plateto the bone. The major disadvantage of these methods is the relative high rate (4-10 precentages) of failure because of the femur head bone which is very brittle and osteoporotic.

This new approach enables the nail a better grip as a result of the cement augmentation which consists of PMMA (Polymethyl methacrylate).

The investigators main goal is to evaluate the use of this surgical technique

ELIGIBILITY:
Inclusion Criteria:

* PFNA augmentation is indicated for severe osteoporotic fractures (Subtrochanteric or intertrochanteric) in the proximal femur.
* Men and women above 80 years old that fuffer from fracture in the proximal femur.

Exclusion Criteria:

* Patient can not come to the follow up clinic visits.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching union at the 3-month and 6-month follow up
  Proportion of patients reaching union at the 3-month and 6-month follow up will be assessed. Union is defined by both clinical evaluation-pain and weight bearing status, and radiological evaluation- three out of four cortices must be bridged as viewed on plain X-ray (AP and lateral views).

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel